CLINICAL TRIAL: NCT03489902
Title: Transvaginal Versus Transobturator Paravaginal Repair Trial
Brief Title: Transvaginal Versus Transobturator Paravaginal Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Ahmed Saaid, Fellow of obstetrics & gynecology, Ain Shams Maternity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVTOPVR
Record Dates: First submitted 2018-03-28; First posted 2018-04-06 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transobturator arm (Experimental): Transobturator Paravaginal Repair
  Interventions: Procedure: Transobturator Paravaginal Repair
- Transvaginal arm (Experimental): traditional transvaginal Paravaginal Repair
  Interventions: Procedure: traditional transvaginal Paravaginal Repair

INTERVENTIONS:
Procedure: Transobturator Paravaginal Repair — Transobturator application of sutures to the white line in cases needing paravaginal repair
  Arms: Transobturator arm
Procedure: traditional transvaginal Paravaginal Repair — traditional transvaginal application of sutures to the white line
  Arms: Transvaginal arm

SUMMARY:
Clinical trial comparing the new technique for paravaginal repair versus the traditional technique

DETAILED DESCRIPTION:
trial comparing the transobturator paravaginal repair versus the traditional technique

ELIGIBILITY:
Inclusion Criteria:

paravaginal defect cystocele

midline and paravaginal defect cystocele

Exclusion Criteria:

* uterine descent previous cystocele surgery

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Operative data | 1 day
  Operative time

SECONDARY OUTCOMES:
Pelvic organ prolapse quantification system | 3 month
  Evaluation of the postoperative degree of anterior vaginal wall descent
Operative Details | 1 day
  blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy HA Saaid, MD, Principal Investigator — Ain Shams University

IPD SHARING:
Plan to Share IPD: No